CLINICAL TRIAL: NCT02622802
Title: Transplacental Transfer of Drugs Used in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Kristel Van Calsteren, MD PhD, Prof Dr, University Hospital, Gasthuisberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PPS201210; 2012-004580-51 (EudraCT Number)
Record Dates: First submitted 2015-06-08; First posted 2015-12-07 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Pregnancy
Keywords: ex-vivo placenta perfusion; transplacental transfer; paracetamol; erythromycin; azithromycin
MeSH Terms: interventions — Acetaminophen; Erythromycin; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ex-vivo placenta perfusion (Experimental): ex vivo placenta perfusion study with exposure to paracetamol, erythromycin and azithromycin
  Interventions: Drug: paracetamol; Drug: Erythromycin; Drug: Azithromycin

INTERVENTIONS:
Drug: paracetamol — In an ex vivo placenta perfusion study, placental tissue is exposed to paracetamol
  Other Names: Paracetamol Sigma Aldrich; acetaminophen
Drug: Erythromycin — In an ex vivo placenta perfusion study, placental tissue is exposed to erythromycin
  Other Names: Erythromycin Sigma Aldrich
Drug: Azithromycin — In an ex vivo placenta perfusion study, placental tissue is exposed to azithromycin
  Other Names: Azithromycin Sigma Aldrich

SUMMARY:
The most important guideline for drug prescription concerning pregnant women is 'drugs should be given only if the maternal benefits outweigh the potential risk to the fetus'. However, poor data is available on maternal drug disposition and transfer through the placenta, so the evidence available for decision making in clinical practice is weak.

An ex-vivo placenta perfusion model will be used to explore the mechanisms governing differences between fetal and maternal drug exposure. The expression of placental transporters and cytochrome P450 (CYP) enzymes will be investigated in primary placenta cell culture and placental biopsies from different gestational stages to learn how the placental drug transfer and disposition is regulated.

The investigators choose to examine the transfer of paracetamol, erythromycin and azithromycin because these drugs are commonly used in human pregnancies and have different metabolic pathways.

DETAILED DESCRIPTION:
1. Background While many drugs are administered to pregnant women, only poor data exist to determine a therapeutically optimal and safe drug treatment in this patient population.

   The general advise on the use of medicines in pregnancy is that you can only prescribe drugs to pregnant women if the benefits for the mother outweigh the risks for the fetus. The problem is that for most medicines safety data are lacking. Most drug effects are dose dependent. So the first step to examine potential fetotoxicity is to test transplacental transfer of drugs.

   Placental transfer from the maternal to the fetal side occurs primarily via passive diffusion, the physicochemical properties of drugs such as lipid solubility, polarity and molecular weight primarily determine the rate of transfer across the placenta. According to membrane permeability properties, low-molecular-weight, lipid-soluble, unbound and unionized compounds can easily cross the human placenta. In addition, some drugs are pumped across the placenta by various active transporters located on both the fetal and maternal side of the trophoblast layer. The most important transporters are P-glycoprotein (P-gp, encoded by the multidrug resistance (MDR)1 gene), Breast cancer resistance protein (BCRP) and multidrug resistance-associated protein (MRP) 1-3 and 5.

   The transfer of foreign chemicals across the placenta can also be modified by metabolism in the placenta itself. The human placenta contains multiple enzyme systems, like CYP2E1 and CYP3A4.
2. Aim & methods:

The aim of this study is to determine fetal drug concentrations of paracetamol, erythromycin and azithromycin by transplacental transport in an ex-vivo placenta perfusion model. Simultaneously collected maternal and fetal drug plasma levels will be compared to assess fetal drug levels based on maternal drug plasma levels.

Moreover, the transporter and metabolizing activity of the trophoblast cells will be examined in a primary human trophoblast culture, and expression of enzymes and transporters will be evaluated at different gestational ages in human placenta biopsies.

Medicines: The investigators choose to examine the transfer of paracetamol, erythromycin and azithromycin because these drugs are commonly used in human pregnancies.

Since the ORACLE trial, erythromycin is in Belgium the first choice treatment in patients with preterm rupture of membranes, despite the fact that the pharmacokinetics (PK) of this drug has been hardly studied in pregnant women. Erythromycin is unstable under acidic conditions while azithromycin is a semi-synthetic macrolide, with a better gastro-intestinal tolerability and tissue penetration than erythromycin and an excellent activity against sexually transmitted pathogens, especially Chlamydia trachomatis. Because of these characteristics more physicians start to switch to azithromycin even without PK data available in pregnancy.

Paracetamol (acetaminophen) is used as first choice painkiller in pregnancy, but also for this drug surprisingly few PK data are available.

ELIGIBILITY:
Inclusion Criteria:

* informed consent has been signed
* (placenta of a) pregnant women with an uncomplicated pregnancy and delivery

Exclusion Criteria:

* use of medication during pregnancy
* hypertension, diabetes
* smoking

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Transplacental transfer rate of drugs and their metabolites measured by comparing the concentrations in simultaneously collected samples from the maternal and fetal compartment in a human ex-vivo placenta perfusion model | 12 months for each drug
  the drug concentrations will be determined by high performance liquid chromatography and mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Kristel Van Calsteren, MD PhD, Principal Investigator — University Hospital Gasthuisberg Leuven
Locations (1):
- University Hospital Gasthuisberg, Leuven, Belgium